CLINICAL TRIAL: NCT04927481
Title: A Multicenter, Open-label, Single-arm, Phase II Study of Mitoxantrone Hydrochloride Liposome Injection in Patients With Advanced HER2 Negative Breast Cancer
Brief Title: A Study of Mitoxantrone Hydrochloride Liposome Injection in Patients With Advanced HER2 Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor has adjusted its R&D strategy.
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE071-CSP-021
Record Dates: First submitted 2021-05-31; First posted 2021-06-16 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitoxantrone Hydrochloride Liposome Injection (Experimental): Patients with advanced HER2 negative breast cancer will receive 20 mg/m2 Mitoxantrone Hydrochloride Liposome injection every 21 days (a cycle) for about 6 cycles.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome Injection

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome Injection — Mitoxantrone Hydrochloride Liposome 20 mg/m2, IV, on day 1 of each 21-day cycle (q3w).

SUMMARY:
This is a multicenter, open-label, single-arm, phase II study to evaluate the safety and efficacy of Mitoxantrone Hydrochloride Liposome in patients with advanced HER2 negative breast cancer.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm, phase II study to evaluate the safety and efficacy of Mitoxantrone Hydrochloride Liposome in patients with advanced HER2 negative breast cancer. Eligible patients will receive Mitoxantrone Hydrochloride Liposome 20 mg/m2 by an intravenous infusion (IV), every 21 days (q3w, 1 cycle) until disease progression, intolerable toxicity, death, or investigator or patient decision.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this study and sign informed consent form;
2. Male or female patients aged 18 to 75 years (inclusive);
3. Histologically confirmed diagnosis of HER-2 negative breast cancer (Including immunohistochemistry HER2 0 or 1+, immunohistochemistry HER2 2+ must be confirmed as negative by in situ hybridization);
4. Patients with unresectable locally advanced or recurrent breast cancer with disease progression after first-line or higher chemotherapy；
5. Hormone receptor (HR) negative breast cancer or HR-positive breast cancer that is not suitable for endocrine treatment or is resistant to endocrine treatment.
6. Prior treatment with both an anthracycline (i.e., doxorubicin or epirubicin) and a taxane (i.e., paclitaxel or docetaxel) at least (acceptable for patients not previously treated with anthracyclines due to high risk factors for cardiotoxicity), and four prior chemotherapy regimens at most；
7. At least one measurable lesion according to RECIST v1.1;
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2;
9. Patients must meet the following criteria prior to treatment (not receiving blood transfusion or growth factors therapy within 14 days before the first administration):

   * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L;
   * Hemoglobin ≥ 90g / L;
   * Platelet count ≥ 90 × 109/L;
   * Creatinine ≤1.5 × upper limit of normal (ULN);
   * Total bilirubin ≤ 1.5×ULN;
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 ×ULN (≤ 5 ×ULN for liver metastasis);
10. For women of childbearing potential: the serum pregnancy test must be negative, and patients are willing to take adequate contraceptive measures during the treatment period and for at least 6 months after the last dose of the study drug;
11. Good compliance and willingness to cooperate with follow-up visits.

Exclusion Criteria:

1. Patients who have severe allergic reactions to mitoxantrone hydrochloride or liposome preparation ingredients;
2. History of other malignancy within 3 years, except for radical cure of carcinoma in situ of the cervix, basal cell carcinoma or squamous cell carcinoma of the skin;
3. Brain metastases and meningeal metastasis;
4. Patients with active hepatitis B (HBsAg positive with hepatitis B virus DNA ≥ 2000 IU/mL), active hepatitis C (hepatitis C virus antibody positive with hepatitis C virus RNA above the lower limit of detection of the study center), or human immunodeficiency virus (HIV) antibody positive;
5. Life expectancy < 3 months;
6. Previous treatment with the anthracyclines, with the total cumulative dose (doxorubicin equivalent) >350 mg/m2;
7. Adverse events from the previous treatment have not resolved to ≤ Grade 1 based on CTCAE (except for the toxicity without safety risk judged by the investigator, such as alopecia, hyperpigmentation);
8. Impaired cardiac function or serious cardiac disease:

   * Long corrected QT interval syndrome or corrected QT interval > 480 ms;
   * Complete left bundle branch block, II-III degree atrioventricular block;
   * Severe, uncontrolled arrhythmias requiring pharmacological treatment;
   * History of chronic congestive heart failure, New York Heart Association ≥ grade 3;
   * Cardiac ejection fraction < 50% within 6 months prior to screening;
   * Heart valve disease with CTCAE ≥ grade 3;
   * ECG evidence of myocardial infarction, unstable angina, severe ventricular arrhythmias, history of severe pericardial disease, and acute ischemic or active conduction system abnormalities within 6 months prior to screening;
9. Uncontrollable hypertension (defined as a measured systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg under pharmacological control);
10. Active bacterial, fungal or viral infections that require intravenous infusion treatment within 1 week prior to the first dose;
11. Any anticancer treatment (including chemotherapy, radiotherapy, molecular targeted therapy, immunotherapy, endocrine therapy) within 4 weeks prior to the first dose, immunomodulators as adjuvant therapy for malignancy within 2 weeks prior to the first dose, any anti-tumor proprietary Chinese medicine (except for those in the category of supporting and relieving symptoms) within 2 weeks prior to the first dose;
12. Patients who enrolled in any other clinical trials within 4 weeks prior to the first dose;
13. Patients who undergone major surgery within 12 weeks before the first dose, or have a surgical schedule during the study period;
14. Patients with thrombosis or thromboembolism within 6 months prior to screening;
15. Lactating female;
16. Serious and/or uncontrolled medical condition that, in the judgment of the investigator, may affect the patient's participation in this study (including, but not limited to: diabetes not effectively controlled, kidney disease requiring dialysis, severe liver disease, life-threatening autoimmune and bleeding disorders, substance abuse, neurological disorders, etc.);
17. Not suitable for this study as decided by the investigator due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From the enrollment to the final documentation of response of the last subject(assessed up to 36 months)
  To investigate the preliminary antitumor efficacy

SECONDARY OUTCOMES:
Disease control rate (DCR) | From the enrollment to the final documentation of response of the last subject(assessed up to 36 months)
  To investigate the preliminary antitumor efficacy
Duration of response (DoR) | From the enrollment to death,lost to follow-up,withdrawal,or study end,whichever occurred first,assessed up to 36 months
  To investigate the preliminary antitumor efficacy
Progression-free survival (PFS) | From the enrollment to death,lost to follow-up,withdrawal,or study end,whichever occurred first,assessed up to 36 months
  To investigate the preliminary antitumor efficacy
Overall survival (OS) | From the enrollment to death,lost to follow-up,withdrawal,or study end,whichever occurred first,assessed up to 36 months
  To investigate the preliminary antitumor efficacy
Treatment emergent adverse events (TEAEs) | from the administration of the first dose to 28 days after the last dose
  The incidence and severity of adverse events, abnormalities in physical exams, vital sign assessments, clinical laboratory assessments, ultrasonic cardiograms (UCGs) and electrocardiographs (ECGs).

CONTACTS AND LOCATIONS:
Overall Officials: qingyuan zhang, PhD, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (29):
- China (29):
  - Anhui Provincial Hospical, Hefei, Anhui
  - Cancer Center Sun Yat-sen University, Guozhou, Guodong
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Daqing People's Hospital, Daqing, Helongjiang
  - Cancer Hospital of Jiamusi City, Jiamusi, Helongjiang
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Cancer Hospital of Henan Province, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhenzhou, Henan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Changsha Kexin Cancer Hospital, Changsha, Hunan
  - Yiyang Central Hospital, Yiyang, Hunan
  - The third Hospital of Nanchang, Nanchang, Jiangxi
  - The second hospital of Jinlin University, Changchun, Jinlin
  - The second hospital of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - The First hospital of China Medical University, Shenyang, Liaoning
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - Sichuan Cancer Hospital & Institute, Chengdu, Sichuan
  - The second people's hospital of neijiang, Neijiang, Sichuan
  - Affiliated tumor Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang